CLINICAL TRIAL: NCT01763684
Title: A Global Comparison of Signature Guides and Conventional Instrumentation in the Oxford Partial Knee
Brief Title: Oxford Signature vs. Conventional Global Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to slow enrollment and not being able to reach the primary endpoint
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO.CR.GK7
Record Dates: First submitted 2012-11-06; First posted 2013-01-09 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee; Osteonecrosis
Keywords: Osteoarthritis; Osteoarthritis, Knee; Osteonecrosis; Arthritis; Knee Arthritis; Knee Replacement
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteonecrosis; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Signature Custom Guides (Active Comparator): Oxford Partial Knee implanted using Signature Custom Guides
  Interventions: Device: Signature Custom Guides
- Conventional Instrumentation (Active Comparator): Oxford Partial Knee implanted using Conventional Instrumentation
  Interventions: Procedure: Conventional Instrumentation

INTERVENTIONS:
Device: Signature Custom Guides — Signature Custom Guides: Signature Custom Guides are intended to be used as a surgical instrument to assist in the positioning of knee replacement components intraoperatively and in guiding the marking of bone before cutting provided that anatomic landmarks necessary for alignment and positioning of the implant are identifiable on patient imaging scans (preoperative MRI).
  Arms: Signature Custom Guides
Procedure: Conventional Instrumentation — Traditional partial knee arthroplasty without the use of Signature technology.
  Arms: Conventional Instrumentation

SUMMARY:
This study will compare alignment criteria in the Oxford Partial Knee using conventional instrumentation and Signature Custom Guides in order to determine if the use of the Signature Custom Guides results in a higher percentage of knees achieving optimal alignment. The study will also examine outcomes with high volume surgeons (>30 cases/year) and low volume surgeons (<10 cases/year).

DETAILED DESCRIPTION:
The primary objectives of this global clinical study are to collect data to assess the following clinical evidence parameters that were gathered from Biomet team members and KOL globally for this product:

1. Evaluate the performance & accuracy of the Oxford Partial Knee System with Signature Knee Guide in comparison to conventional instrumentation.
2. Compare the accuracy of Signature Guides between two user profiles: high volume surgeons & low volume surgeons in a global mix.
3. Assess potential economic & efficiency advantages in the short term and long-term: OR efficiency, patient quality of life and activity, clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Intended for use in individuals with osteoarthritis or Avascular necrosis limited to the medial compartment of the knee that is also lacking patellofemoral or lateral compartment disease.
* Use of cementless femoral fixation is permitted outside of the United States if it complies with all local, state, and/or national and international regulations. The same technique must be used consistently throughout the course of the study with all cases
* Patients 21 and over

Exclusion Criteria:

* Use of Cementless Fixation in the United States
* Infection, sepsis or osteomyelitis
* Use in lateral compartment of the knee
* Rheumatoid arthritis or other forms of inflammatory joint disease
* Revision of failed prosthesis, failed upper tibial osteotomy, or post traumatic arthritis after tibial plateau fracture
* Insufficiency of the collateral, anterior, or posterior cruciate ligaments which would preclude stability of the device.
* Disease or damage to the lateral compartment of the knee
* Uncooperative patient or patient with neurologic disorders who is incapable of following directions
* Osteoporosis in the United States / Insufficient bone stock outside the United States
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to implant site
* Rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, neuromuscular disease.
* Incomplete or deficient soft tissue surrounding the knee.
* Charcot's disease
* A fixed varus deformity (not passively correctable) of greater than 15 degrees
* A flexion deformity greater than 15 degrees.
* Non-staged Bilateral patients
* Patients who refuse, cannot, or should not receive a CT or MRI. Since patients are randomized into treatment groups, all patients must be able to receive an MRI (should follow local MRI screening protocol). This excludes patients who have metal artifacts in the knee, patients who are too large to fit into the knee coil, patients with pacemakers, patients unable to lie still for the duration of the MRI, and patients who are claustrophobic.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schenck, Ph.D., Study Director — Zimmer Biomet
Locations (7):
- United States (7):
  - Orthopedic and Sports Medicine Center, Elkhart, Indiana
  - The Orthopaedic Center, Rockville, Maryland
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Joint Implant Surgeons, Columbus, Ohio
  - Texas Institute for Hip & Knee Surgery, Austin, Texas
  - Advanced Orthopedics, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Bi-lateral treatment was not recorded. Each treated knee is counted as 1 participant.
Period: Overall Study
Arm/Group | Signature Custom Guides | Conventional Instrumentation
Started | 133 | 133
Completed Surgery | 126 | 127
Completed | 0 | 0
Not Completed | 133 | 133
Not completed — Study terminated early due to low enrollment | 126 | 127
Not completed — Study surgery not performed | 7 | 6

BASELINE CHARACTERISTICS:
Population: All patients that completed the index surgery. Bilateral treatment was not recorded, all patients are counted as 1 treated knee.
Groups:
- Total: Total of all reporting groups
Arm/Group | Signature Custom Guides | Conventional Instrumentation | Total
Number analyzed (Participants) | 126 | 127 | 253
Age, Categorical [Count of Participants; unit: Participants] — Population: 5 patients age not reported
  Participants
    number analyzed (Participants) | 122 | 126 | 248
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 77 | 77 | 154
    >=65 years | 45 | 49 | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: 5 patient conventional age missing
  Years
    number analyzed (Participants) | 126 | 122 | 248
    (all) | 63.2 (10.0) | 62.5 (9.1) | 62.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 5 patients gender not reported
  Participants
    number analyzed (Participants) | 126 | 122 | 248
    Female | 56 | 68 | 124
    Male | 70 | 54 | 124
Region of Enrollment [Number; unit: participants] — Population: 5 subjects no region data available
  participants
    United States: number analyzed (Participants) | 126 | 122 | 248
    United States | 95 | 71 | 166
    Europe: number analyzed (Participants) | 126 | 122 | 248
    Europe | 25 | 47 | 72
    Australia: number analyzed (Participants) | 126 | 122 | 248
    Australia | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Knees Achieving Optimal Alignment
Description: Percentage of Knees Achieving Optimal Alignment defined as a difference of 5 or less between all target and observed angles.
Time Frame: 12 weeks
Population: Data from all patients as treated
Measure: Number; unit: percentage of total
Arm/Group | Signature Custom Guides | Conventional Instrumentation
Number analyzed (Participants) | 100 | 94
percentage of total | 45 | 29

2. Secondary Outcome: Instruments Used During Surgery
Description: Number of Instrument cases used to complete index surgery.
Time Frame: Operative
Population: All patients as treated
Measure: Mean (Standard Deviation); unit: Instrument cases
Arm/Group | Signature Custom Guides | Conventional Instrumentation
Number analyzed (Participants) | 122 | 126
Instrument cases | 4.2 (0.76) | 3.8 (0.97)

3. Secondary Outcome: Knee Society Functional Score
Description: Functional Score from Knee Society Score. These are 3 of the 10 items. Scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions
Time Frame: 1 Year
Population: All patients, as treated, reaching the 1 year follow up datapoint with Knee Society Score score completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Signature Custom Guides | Conventional Instrumentation
Number analyzed (Participants) | 58 | 60
units on a scale | 88.1 (18.2) | 91.8 (14.2)

4. Secondary Outcome: Leg Alignment Femoral Varus/Valgus
Description: Mechanical Leg Alignment of Components (degrees): Difference of Femoral Varus/Valgus angle as measured via CT-scan directly post-operative, vs target angle
Time Frame: Directly Postoperative
Population: All patients as treated with post-operative CT collected
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Signature Custom Guides | Conventional Instrumentation
Number analyzed (Participants) | 100 | 94
Degrees | 3.55 (2.7) | 4.75 (3.53)

5. Secondary Outcome: Blood Loss
Description: Blood Loss during surgery
Time Frame: Right after surgery (up to 2 hours after surgery)
Population: All patients as treated for which blood loss is recorded
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Signature Custom Guides | Conventional Instrumentation
Number analyzed (Participants) | 49 | 79
ml | 81.9 (84.5) | 54.8 (73.0)

6. Secondary Outcome: Knee Society Objective Score
Description: Objective score from Knee Society Score. These are 7 of the 10 items. Scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions
Time Frame: 1 Year
Population: All patients, as treated, reaching the 1 year follow up datapoint with Knee Society Score completed
Measure: Mean (Standard Deviation); unit: units on a scale from 0 to 100
Arm/Group | Signature Custom Guides | Conventional Instrumentation
Number analyzed (Participants) | 58 | 60
units on a scale from 0 to 100 | 93.3 (16.3) | 95.0 (17.5)

7. Secondary Outcome: Oxford Knee Score
Description: Oxford Knee Score (OKS). Scored from 0 to 48 with 0 being the worst possible outcome and 48 being the best outcome
Time Frame: 1 Year
Population: All patients, as treated, reaching the 1 year follow up datapoint with Oxford Knee Score completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Signature Custom Guides | Conventional Instrumentation
Number analyzed (Participants) | 58 | 57
units on a scale | 42.6 (6.1) | 44.0 (4.9)

8. Secondary Outcome: EQ5D Score
Description: EuroQol 5D Quality of Life score. Range from 0 to 1 with 1 being the best outcome.
Time Frame: 1 Year
Population: All patients, as treated, reaching the 1 year follow up datapoint with EQ5D score completed
Measure: Mean (Standard Deviation); unit: units on a scale from 0 to 1
Arm/Group | Signature Custom Guides | Conventional Instrumentation
Number analyzed (Participants) | 58 | 58
units on a scale from 0 to 1 | 0.88 (0.15) | 0.9 (0.19)

9. Secondary Outcome: Leg Alignment Femoral Flexion/Extension
Description: Mechanical Leg Alignment of Components (degrees): Difference of Femoral Flexion/Extension angle as measured via CT-scan directly post-operative, vs target angle
Time Frame: Directly Postoperative
Population: All patients as treated with post-operative CT collected
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Signature Custom Guides | Conventional Instrumentation
Number analyzed (Participants) | 89 | 88
Degrees | 3.48 (2.7) | 4.59 (3.34)

10. Secondary Outcome: Leg Alignment Tibial Varus/Valgus
Description: Mechanical Leg Alignment of Components (degrees): Difference of Tibial Varus/Valgus angle as measured via CT-scan directly post-operative, vs target angle
Time Frame: Directly Postoperative
Population: All patients as treated with post-operative CT collected
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Signature Custom Guides | Conventional Instrumentation
Number analyzed (Participants) | 100 | 91
Degrees | 4.04 (2.41) | 4.10 (2.39)

11. Secondary Outcome: Leg Alignment Tibial Flexion/Extension
Description: Mechanical Leg Alignment of Components (degrees): Difference of Tibial Flexion/Extension angle as measured via CT-scan directly post-operative, vs target angle
Time Frame: Directly Postoperative
Population: All patients as treated with post-operative CT collected
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Signature Custom Guides | Conventional Instrumentation
Number analyzed (Participants) | 94 | 100
Degrees | 2.47 (2.06) | 2.96 (2.04)

ADVERSE EVENTS:
Arm/Group | Signature Custom Guides | Conventional Instrumentation
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/133
Serious Adverse Events (participants affected / at risk) | 3/133 | 6/133
Other Adverse Events (participants affected / at risk) | 12/133 | 18/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Signature Custom Guides (N=133) | Conventional Instrumentation (N=133)
PERFORATED DIVERTICULITIS, HINCHEY IV (Gastrointestinal disorders) | 0 (0) | 1 (1)
DEHISCENCE OF PROXIMAL MEDIAL CAPSULAR SUTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LAPARAOSCIPIC GASTRIC BYPASS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ARTHROSCOPIC PROCEDURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — PAIN AND SWELLING DUE TO LOOSE BODY RESULTING IN OUTPATIENT ARTHROSCOPIC PROCEDURE. SYNOVITIS, SMALL LATERAL MENISCAL TEAR AND PIECE OF CEMENT WERE IDENTIFIED AND REMOVED. PATIENT WENT HOME THE SAME DAY
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — PAIN LEFT SHOULDER RESULTING IN SHOULDER SURGERY ON 6 OCT 2014 (IMPINGEMENT SYNDROME AND ACROMIOCLAVICULAR ARTHRITIS)
Patient Fall (General disorders) | 0 (0) | 1 (1) — PATIENT FELL GETTING OUT OF BED DUE TO LEG NUMBNESS FROM BL SOCIAL ADMISSION TO HOSPITAL BECAUSE FALL AND NUMBNESS. SLIPPED OUT OF BED.
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — PERSISTANT PAIN PROBLEM RIGHT KNEE
Knee Gonarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — TOTAL KNEE PROSTHESIS Contralateral ON 27 FEB 2015 DUE TO MEDIAL GONARTHROSIS LEFT
Unkown event (General disorders) | 0 (0) | 1 (1) — Unknown description
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Signature Custom Guides (N=133) | Conventional Instrumentation (N=133)
2 MM BLOOD BLISTER ON INCISION ON OPERATIVE KNEE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — 2 MM BLOOD BLISTER ON INCISION ON OPERATIVE KNEE
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
DEGENERATIVE DISC DISEASE LUMBAR SPINE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
DELAYED WOUND HEALING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — DELAYED WOUND HEALING
Disease Progression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — LATERAL COMPARTMENT DISEASE PROGRESSION
Fall (General disorders) | 0 (0) | 1 (1) — PATIENT FALLS ON HIS KNEE
FEELING OF RIGHT KNEE GIVING WAY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Knee popping/clicking (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Knee Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — Postoperative swelling
PATELLA TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
POST-OP NAUSEA (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No